CLINICAL TRIAL: NCT02579291
Title: Changes in Spasticity, Motor Function and Stabilometry After Dry Needling of the Tibialis Posterior Muscle in Post-stroke Patients
Brief Title: Dry Needling in Patients Who Had Experience Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC 07-2015
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: Stroke; Dry needling; Spasticity; Motor function; Stabilometry
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dry needling (Experimental): The experimental group will receive a single session of Bobath therapy including techniques targeting modulation of central nervous system. In addition, this group will receive a single session of dry needling into the tibialis posterior muscle with a disposable stainless steel needle (0.3mm x 50mm)
  Interventions: Other: Dry needling
- Bobath (Active Comparator): This group will receive a single session of Bobath therapy including techniques targeting modulation of central nervous system.
  Interventions: Other: Bobath

INTERVENTIONS:
Other: Dry needling — Once the most painful spot is located within a palpable spastic taut band, the overlying skin is cleaned with alcohol. The needle will be inserted, penetrating the skin about 15-20mm, until the first local twitch response is obtained. Once the first local twitch response is obtained, the needle will be moved up and down (4 to 5 mm. vertical motions with no rotation) in the muscle at approximately 1Hz for 25-30 seconds.
  Arms: Dry needling
Other: Bobath — Patients will receive different neuromodulatory interventions based on the Bobath concept with the aim to decrease spasticity on the lower extremity
  Arms: Bobath

SUMMARY:
Individuals who had experience a stroke usually suffer from spasticity at medium and long-terms. The presence of spasticity in the lower extremity implies several impairments for standing and walking inducing high disability. A recent study has proposed the use of dry needling for improving spasticity in the lower extremity. No study has investigated the effects of deep dry needling inserted into spastic musculature in stabilometry and moto function in patients who had experience a stroke. A randomized controlled trial investigating the effects of the inclusion of deep dry needling into a Bobath interventional program on spasticity, motor function and balance (stabilometry) in individuals who had experience a stroke

ELIGIBILITY:
Inclusion Criteria:

* First-ever unilateral stroke;
* hemiplegia resulting from stroke;
* unilateral equinovarus gait with independent walk;
* able to ambulate without supporting devices

Exclusion Criteria:

* recurrent stroke;
* previous treatment with nerve blocks, motor point injections with neurolytic agents for spasticity at any time, or with BTX-A in the previous 6 months
* not independent in the basic activities of daily living
* cognitive deficits;
* progressive or severe neurologic diseases;
* fear to needles;
* any contraindication for dry needling

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in spasticity before and 10 minutes after the intervention | Baseline and immediate after the intervention
  Spasticity in the affected ankle joint will be evaluated with the Modified Modified Ashworth Scale (MMAS). The examiner passively will move the ankle in dorsal-flexion direction, back and forth at least 5 times and will evaluate the degree of resistance to the movement on a scale from 0-4.

SECONDARY OUTCOMES:
Changes in motor function before and 10 minutes after the intervention | Baseline and immediate after the intervention
  The Fugl-Meyer evaluation will be used to determine motor impairments and physical recovery of patients who had experienced a stroke
Changes in stabilometry outcomes before and 10 minutes after the intervention | Baseline and immediate after the intervention
  The time reaction will be assessed as stabilometric data from each patient.

CONTACTS AND LOCATIONS:
Overall Officials: CESAR FERNANDEZ-DE-LAS-PEÑAS, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Cesar Fernandez-de-Las-Peñas, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Sanchez-Mila Z, Salom-Moreno J, Fernandez-de-Las-Penas C. Effects of dry needling on post-stroke spasticity, motor function and stability limits: a randomised clinical trial. Acupunct Med. 2018 Dec;36(6):358-366. doi: 10.1136/acupmed-2017-011568. Epub 2018 Jul 9. PMID 29986902